CLINICAL TRIAL: NCT02831036
Title: The Impact of Physical Exercise on Navigation Performance in Soldier
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Bar-Ilan University, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SHEBA-16-3321-HS-CTIL
Record Dates: First submitted 2016-07-10; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Spatial Learning
MeSH Terms: conditions — Spatial Learning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- trial group (Experimental): subjects in trial group will be following the experimental protocol (VO2max tests and spatial orientation tests) while performing a training program during the trial (3 months).
  Interventions: Other: training program; Other: VO2max test; Other: spatial orientation test
- control group (Other): following the experimental protocol (VO2max tests and spatial orientation tests)without performing additional exercise.
  Interventions: Other: VO2max test; Other: spatial orientation test

INTERVENTIONS:
Other: training program — subjects in the trial group will follow a training program which includes 3 times a week running on a treadmill.
  Arms: trial group
Other: VO2max test — each subject will perform 4 times VO2max test according to BRUCE protocol in order to evaluate his aerobic fitness.
Other: spatial orientation test — each subject will undergo 4 spatial orientation tests during the trial (month between 2 tests), each test is composed of 5 following days in which the subject will wear virtual reality glasses (Oculus Rift DK2) and attempt to arrive different destinations in a virtual maze tasks (using xbox one controller). each day will be given 3 attempts, the duration of each attempt is 2 min.

SUMMARY:
20 healthy man, 10 in trial group and 10 in control group (randomly divided) will participate in the experiment on order to evaluate if improvement in physical fitness influences spatial learning in humans.

DETAILED DESCRIPTION:
subjects in both groups will perform 4 sets of VO2max test and spatial orientation test with a month between them (total 3 month).

in addition, subjects in trial group will follow a training program throughout the trial (running on treadmill 3 times a week), suited according to their result in the first VO2max test.

in each set VO2max test will be perform before spatial orientation test , in order to evaluated the subject's aerobic fitness. the spatial orientation test is composed of 5 following days in which the subject has 3 attempts to arrive to a destination in xbox one controller using a virtual glasses (Oculus Rift DK2). each attempt duration is 2 min.

ELIGIBILITY:
Inclusion Criteria:

* civilian healthy man, aged 18-30
* without any neurological or psychiatric disorder
* not wearing eyeglasses

Exclusion Criteria:

* athletes or trained man (for both groups)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
spatial learning (composite) | 20 experimental days for each participant
  each spatial orientation test length is 5 days. spatial learning is evaluated through time for completion and number of errors out of 3 attempts each day.

SECONDARY OUTCOMES:
maximal aerobic capacity | 4 experimental days for each participant
  VO2max tests along the trial are performed in order to evaluate the improvement or lack of improvement in both groups in correlation with their spatial learning.

CONTACTS AND LOCATIONS:
Overall Officials: Haggai Schermann, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Ramat- Gan, Israel

IPD SHARING:
Plan to Share IPD: No